CLINICAL TRIAL: NCT00722397
Title: Studies to Treat Or Prevent Pediatric Type 2 Diabetes (STOPP-T2D) Treatment Options for Type 2 Diabetes in Adolescents and Youth (TODAY) Genetics Study
Brief Title: TODAY Genetics Study
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: IND - DK61230-GENETICS; DK61230
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes
Keywords: genetics, pediatrics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Collect 27 mL of blood to send (1) for extraction of DNA to the NIDDK Central Repository and (2) for measurement of glucose, C-peptide, and autoantibody analysis to a central blood laboratory.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The TODAY study group has prepared a protocol with the primary objective of collecting blood and phenotypic information to be used to explore relationships between candidate genes and type 2 diabetes (T2D), as well as obesity, insulin resistance, and cardiovascular complications of insulin resistance. Participation in the genetics study includes a blood draw for analysis of diabetes type and DNA extraction, as well as collection of basic family and medical history. Appropriate informed consent and assent are obtained from all participants to extract DNA and send blood, genetic material, and medical history to the Central Repository of the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) of the National Institutes of Health (NIH). The data are kept indefinitely by the Central Repository. The NIDDK will issue requests for proposals (RFP) throughout the scientific community for research that may help in the development of new diagnostic tests, new treatments, and new ways to prevent diabetes and other related comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes by ADA criteria (laboratory determinations of fasting glucose ≥ 126 mg/dL, random glucose ≥ 200 mg/dL, or two-hour oral glucose tolerance test (OGTT) glucose ≥ 200 mg/dL) documented and confirmed in medical record or a laboratory determination of HbA1c ≥ 7%. For asymptomatic patients diagnosed with diabetes with a normal fasting glucose but an elevated two-hour glucose during an OGTT, the HbA1c must be ≥ 6%.
* BMI ≥ 85th percentile documented at time of diagnosis or at screening.
* Age < 18 at time of diagnosis.
* Signed informed consent and assent forms as appropriate.

Exclusion Criteria:

* Genetic syndrome or disorder known to affect glucose tolerance other than diabetes.
* Patient on medication known to affect glucose tolerance, insulin sensitivity or secretion within 60 days of the time of diagnosis. If diagnosis is confirmed after the patient has been off the medication for 60 days, the patient may be included. Exclusionary medications include but are not limited to

  1. inhaled steroids at dose above 1000 mcg daily fluticasone equivalent,
  2. oral glucocorticoids,
  3. antirejection or chemotherapy agents (e.g., tacrolimus, L-asparaginase),
  4. atypical antipsychotics.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment is conducted within a 'catchment' area that includes (a) the patient pools of the 15 TODAY clinical centers and (b) collaborating clinics and physicians who either refer subjects to a TODAY site or obtain IRB approval to conduct the protocol at their own locale.
Sampling Method: Probability Sample
Enrollment: 2654 (Actual)
Dates: Start 2008-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Blood draw to be processed and analyzed to yield genetic data. | Blood is drawn at the single study visit.
  Blood is sent to the DNA processing center identified by NIDDK for processing and shipment to the NIDDK Repository.

SECONDARY OUTCOMES:
Phenotype data. | Collected at single study visit.
  Demographic, medical history, and other data about participant and family, by self-report.
Laboratory values. | Single study visit.
  Serum glucose, C-peptide, and pancreatic autoimmunity antibodies determined by study central laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Zeitler, MD PhD, Principal Investigator — University of Colorado, Denver; Kathryn Hirst, PhD, Principal Investigator — George Washington University
Locations (25):
- United States (25):
  - UAMS Arkansas Children's Hospital, Little Rock, Arkansas
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCSD Rady Children's Hospital, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - George Washington University Biostatistics Center, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Kansas City Children's Mercy Hospital, Kansas City, Missouri
  - St Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- [Result] Srinivasan S, Chen L, Todd J, Divers J, Gidding S, Chernausek S, Gubitosi-Klug RA, Kelsey MM, Shah R, Black MH, Wagenknecht LE, Manning A, Flannick J, Imperatore G, Mercader JM, Dabelea D, Florez JC; ProDiGY Consortium. The First Genome-Wide Association Study for Type 2 Diabetes in Youth: The Progress in Diabetes Genetics in Youth (ProDiGY) Consortium. Diabetes. 2021 Apr;70(4):996-1005. doi: 10.2337/db20-0443. Epub 2021 Jan 21. PMID 33479058